CLINICAL TRIAL: NCT03667716
Title: A Phase 1a/1b Study of COM701 as Monotherapy and In Combination With an Anti-PD-1 Antibody in Subjects With Advanced Solid Tumors.
Brief Title: COM701 (an Inhibitor of PVRIG) in Subjects With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Compugen Ltd (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPG-01-001
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Advanced Cancer; Ovarian Cancer; Breast Cancer; Lung Cancer; Endometrial Cancer; Ovarian Neoplasm; Triple Negative Breast Cancer; Lung Neoplasm; Neoplasm Malignant; Colo-rectal Cancer
Keywords: PVRIG; advanced cancer; checkpoint inhibitor; DNAM (DNAX Accessory molecule 1); PD-1 inhibitor; CD112; CD 112R; Poliovirus receptor-related immunoglobulin; PVRL2; Nivolumab; opdivo; TIGIT antibody; COM902
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Lung Neoplasms; Endometrial Neoplasms; Triple Negative Breast Neoplasms; Neoplasms; Colonic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- P1a Arm A (Monotherapy Dose Escalation). (Experimental): COM701 monotherapy sequential dose escalation administered IV every 3 weeks and a Cohort IV every 4 weeks. Up to 8 dose escalation cohorts may be evaluated until a maximum tolerated dose or recommended phase 2 dose is identified.
  Interventions: Drug: COM701
- P1a Arm B (Combination Dose Escalation). (Experimental): COM701 sequential dose escalation administered IV every 3 weeks in combination with Opdivo (Nivolumab) 360mg administered IV every 3 weeks and COM701 administered IV every 4 weeks in combination with Opdivo (Nivolumab) 480mg administered IV every 4 weeks.
  Interventions: Drug: COM701 with Opdivo (Nivolumab).
- P1a Arm A (Monotherapy Expansion). (Experimental): COM701 monotherapy administered IV every 4 weeks. Cohort expansion in subjects with the following select tumor types (NSCLC, Breast, Ovarian, Endometrial and Colorectal cancer).
  Interventions: Drug: COM701
- P1b (Combination Cohort Dose Expansion). (Experimental): COM701 administered IV every 4 weeks in combination with Opdivo (Nivolumab) 480 mg administered IV every 4 weeks. Cohort expansion in subjects with the following select tumor types (Breast, Ovarian, Endometrial and Colorectal cancer).
  Interventions: Drug: COM701 with Opdivo (Nivolumab).

INTERVENTIONS:
Drug: COM701 — COM701 monotherapy.
  Arms: P1a Arm A (Monotherapy Dose Escalation).; P1a Arm A (Monotherapy Expansion).
Drug: COM701 with Opdivo (Nivolumab). — COM701 in combination with Opdivo (Nivolumab).
  Arms: P1a Arm B (Combination Dose Escalation).; P1b (Combination Cohort Dose Expansion).

SUMMARY:
This is a Phase 1 open label sequential dose escalation and cohort expansion study evaluating the safety, tolerability and preliminary clinical activity of COM701 as monotherapy and in combination with nivolumab.

DETAILED DESCRIPTION:
This Phase 1 study evaluates the safety, tolerability, Pharmacokinetics (PK) and preliminary clinical activity of COM701 an inhibitor of poliovirus receptor related immunoglobulin domain containing (PVRIG) as monotherapy and in combination with nivolumab in subjects with advanced solid tumors. Cohort expansion will be explored evaluating COM701 monotherapy and in combination with nivolumab in subjects with the following select tumor types (Non-Small cell lung cancer (NSCLC), Ovarian, Breast (including Triple negative breast cancer (TNBC) and endometrial cancer. Other tumor types such as CRC-MSS, CRC-KRAS mutant will be enrolled based on emerging clinical activity data.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Subjects who received prior immune-stimulatory antitumor agents, such as anti-PD-1, anti-PD-L1, anti-CTLA-4, OX-40, CD137, etc. are eligible.
* Histologically or cytologically confirmed, locally advanced or metastatic solid malignancy and has exhausted all the available standard therapy or is not a candidate for the available standard therapy.

Select Tumor Types (COM701 monotherapy cohort expansion; COM701 in combination with nivolumab):

* Breast cancer (TNBC): Histologically confirmed incurable, advanced estrogen receptor-, progesterone receptor-, and human epidermal growth factor receptor 2 (HER2)-negative (triple-negative) adenocarcinoma of the breast, as defined by the American Society of Clinical Oncology-College of American Pathologists (ASCO-CAP) guidelines. Disease recurrence or progression during or after at least one systemic treatment that included an anthracycline and/or a taxane in the neoadjuvant, adjuvant, or metastatic setting. Subjects must have progressed after a poly ADP-ribose polymerase (PARP) inhibitor for patients with deleterious or suspected deleterious germline breast cancer susceptibility gene (BRCA) mutated metastatic breast cancer. P1b COM701 + nivolumab expansion cohort, COM701 monotherapy expansion cohort.
* Endometrial cancer: Subjects with locally advanced or metastatic endometrial cancer, disease recurrence or progression during or after prior therapy that included platinum-based chemotherapy. P1b COM701 + nivolumab expansion cohort, COM701 monotherapy expansion cohort.
* Ovarian cancer: Disease recurrence or progression during or after prior therapy that included: surgical resection, platinum agent, PARP inhibitor (for subjects with deleterious or suspected deleterious germline BRCA-mutated advanced ovarian cancer or as a maintenance therapy for subjects who have had complete or partial response to platinum-based therapy). P1b COM701 + nivolumab expansion cohort, COM701 monotherapy expansion cohort.
* NSCLC: Documented stage IIIB or IV or recurrent NSCLC, Disease recurrence or progression during or after prior treatment that included: platinum agent, targeted therapy such as a TKI (if with biopsy-confirmed cytogenetic mutation eg EGFR, ROS, BRAF). COM701 monotherapy expansion cohort.
* CRC (microsatellite stable, KRAS mutation) - P1b COM701 + nivolumab expansion cohort, COM701 monotherapy expansion cohort.
* For Phase 1a monotherapy expansion and Phase 1b only: subject has at least one measurable lesion that could be followed during the study according to RECIST v1.1.

Key Exclusion Criteria:

* Active autoimmune disease requiring systemic therapy in the last 2 years prior to the first dose of COM701.
* Symptomatic interstitial lung disease or inflammatory pneumonitis.
* History of immune-related events that lead to immunotherapy treatment discontinuation.
* Untreated or symptomatic central nervous system (CNS) metastases.
* Impaired cardiac function or clinically significant cardiac disease, including any of the following: a) Unstable angina pectoris ≤ 6 months prior to first scheduled dose of COM701; b) Acute myocardial infarction ≤ 6 months prior to first scheduled dose of COM701.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of subjects with Adverse Events (AEs) as per CTCAE v4.03 and Dose-Limiting Toxicities (DLTs). | DLT evaluation window in the 1st cycle (21 or 28 days).
  To evaluate the safety profile of COM701 monotherapy and in combination with nivolumab.
Determine the maximum tolerated dose (MTD) and/or the recommended dose for expansion (RDFE) (COM701 monotherapy and in combination with nivolumab). | Approximately 2 year.

SECONDARY OUTCOMES:
Incidence of subjects with Anti-COM701 antibody. | Approximately 2 years.
  Immunogenicity of COM701 monotherapy and in combination with nivolumab.
Overall Response Rate as per RECIST v1.1 | Approximately 2 years.
  Preliminary antitumor activity of COM701 in combination with nivolumab.

CONTACTS AND LOCATIONS:
Overall Officials: COM701 Study Director, Study Director — Compugen USA, Inc.
Locations (11):
- United States (11):
  - University of California Los Angeles (UCLA)., Los Angeles, California
  - Florida Cancer Specialists, Sarasota, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest., Grand Rapids, Michigan
  - Columbia University, New York, New York
  - Cleveland Clinic., Cleveland, Ohio
  - The University of Tennessee WEST Cancer Center., Memphis, Tennessee
  - Sarah Cannon Research Institute., Nashville, Tennessee
  - M D Anderson Cancer Center., Houston, Texas
  - The START Center for Cancer Care., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No